CLINICAL TRIAL: NCT06841887
Title: Unlock the Power of Resona 9 Ultrasound Machine: an Observational Study to Set-up and Test New Advanced Vascular Imaging Protocols
Brief Title: New Advanced Vascular Imaging Ultrasound Protocols
Acronym: RESONA-SETTING
Status: Recruiting | Type: Observational
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: RESONA-SETTING
Record Dates: First submitted 2025-02-03; First posted 2025-02-24 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Renal Diseases; Cerebral Disorder
Keywords: ultrasound; imaging; vascular protocol
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Males, age group 1: Male subjects aged 18-40 years
  Interventions: Diagnostic Test: US acquisitions
- Males, age group 2: Male subjects aged 41-55 years
  Interventions: Diagnostic Test: US acquisitions
- Males, age group 3: Male subjects aged 56-75 years
  Interventions: Diagnostic Test: US acquisitions
- Female, age group 1: Female subjects aged 18-40 years
  Interventions: Diagnostic Test: US acquisitions
- Females, age group 2: Female subjects aged 41-55 years
  Interventions: Diagnostic Test: US acquisitions
- Females, age group 3: Female subjects aged 56-75 years
  Interventions: Diagnostic Test: US acquisitions

INTERVENTIONS:
Diagnostic Test: US acquisitions — US acquisition from two anatomical regions i.e., the non-dominant arm and the neck.

SUMMARY:
This is a single-center observational study aimed at setting up and testing new ultrasound vascular imaging protocols, conducted exclusively for research purposes. The study will perform US examinations in 60 subjects. The subjects enrolled in the study will be examined the first time and will then provide consent to be examined again in the future if needed.

The primary aim of this study is to set-up and test new advanced US protocol for the arm and cerebral blood vessels

The secondary objectives will be:

* Define ranges of normality/reference values of US-based parameters to be compared with pathological values.
* Evaluate the repeatability and reproducibility of the acquired US measurements.
* Evaluate the correlation between age and the acquired US measurements.
* Evaluate the correlation between gender and the acquired US measurements.

DETAILED DESCRIPTION:
The Medical Imaging Laboratory of Istituto di Ricerche Farmacologiche Mario Negri IRCCS deals with the processing of diagnostic images, allowing quantitative analysis of anatomical structures and organs functions in vivo. The research activities of the group are focused on: i) developing novel techniques to segment and quantify anatomical structures and pathological lesions in response to specific clinical needs; ii) identifying and validating novel imaging biomarkers, iii) investigating novel morphologic and hemodynamic changes in different vascular districts and the role of hemodynamics in vascular disease onset and progression. Besides these activities, increasing efforts have recently been devoted to exploring the potential of novel imaging solutions and in setting up new non-invasive imaging protocols. These protocols have been primarily developed for the kidney and renal arteries, the cerebral vasculature, and the arteriovenous fistula used in hemodialysis, which are the main focus of the Medical Imaging Lab's activities. Specifically, in 2024 Istituto di Ricerche Farmacologiche Mario Negri IRCCS purchased the new ultrasound (US) machine Resona 9, within the ANTHEM project (ID: NCT05996731). Resona 9 is the top-of-the-line model among Mindray's ultrasound machines. It combines advanced features to deliver exceptional image quality with a suite of artificial intelligence-enhanced technologies designed to help clinicians improve reproducibility and optimize productivity. Specifically related to our research focus, the Resona 9 incorporates novel advanced functionalities to accurately measure vascular wall thickness and stiffness. Moreover, the VFlow technique enables the visualization of complex blood flow features. Our Resona 9 is also equipped with the PIUR tUS device, which transforms the US system into a tomographic 3D solution device. This allows the acquisition of a stack of images of the blood vessels and the reconstruction of 3D virtual models, with big advantages in terms of costs and velocity of the acquisition as compared to conventional magnetic resonance imaging.

To take full advantage of all these US-based techniques and make the most out of Resona 9 tools on patients with renal and cerebral pathologies, there is an urgent need of setting up dedicated US protocols and testing. This step will also allow collecting ranges of normality/reference values of image-based parameters, to be later used to compare with corresponding specific parameters acquired in patients.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Female and/or male aged between 18 and 75 years
* No previous history of kidney or cerebral disease and no pathologies that might have affected the vascular system

Exclusion Criteria:

* Previous history of kidney or cerebral disease or pathologies that might have affected the vascular system
* Legal incapacity, limited legal capacity, intellectual disability, uncooperative attitude or any other evidence that the subject will not be able to understand the study aims and procedures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participation in this study will be proposed to subjects with no previous history of kidney or cerebral disease, and no pathologies that might have affected the vascular system (hypertension, diabetes). Sixty subjects will be studied, 30 females and 30 males. For both genders, they must be equally distributed within 3 age-groups: 18-40 years, 41-55 years and 56-75 years.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Non-dominant arm US acquisitions | US acquisition at enrollment
  Diameter of the radial artery in the middle forearm, brachial artery over the elbow, ulnar artery in the middle forearm and Cephalic vein in the middle forearm (mm)
Non-dominant arm US acquisitions | US acquisition at enrollment
  Flow volume of the radial artery in the middle forearm, brachial artery over the elbow, ulnar artery in the middle forearm (ml/min)
Non-dominant arm US acquisitions | US acquisition at enrollment
  Thickness of the radial artery and cephalic vein wall (mm)
Non-dominant arm US acquisitions | US acquisition at enrollment
  Stiffness of the radial artery and cephalic vein wall (%)
Non-dominant arm US acquisitions | US acquisition at enrollment
  Time averaged velocity (TAV) of the radial artery in the middle forearm, brachial artery over the elbow and ulnar artery in the middle forearm (cm/s)
Neck carotid (right and left) US acquisitions | US acquisition at enrollment
  Diameter of the common carotid artery, internal carotid artery, external carotid artery and vertebral arteries (mm)
Neck carotid (right and left) US acquisitions | US acquisition at enrollment
  Flow volume of the common carotid artery, internal carotid artery, external carotid artery and vertebral arteries (ml/min)
Neck carotid (right and left) US acquisitions | US acquisition at enrollment
  Thickness of the wall of the common carotid (mm)
Neck carotid (right and left) US acquisitions | US acquisition at enrollment
  Stiffness of the wall of the common carotid (%)
Neck carotid (right and left) US acquisitions | US acquisition at enrollment
  Time averaged velocity (TAV) of the common carotid artery, internal carotid artery, external carotid artery and vertebral arteries (cm/s)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, M.D., Study Director — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (1):
- Clinical Research Centre for Rare Diseases Aldo e Cele Daccò, Ranica, BG, Italy

IPD SHARING:
Plan to Share IPD: Undecided